CLINICAL TRIAL: NCT05983380
Title: The Effect of Hand Mobility and Grip Strengthening Exercises on Upper Limb Volume, Quality of Life, and Hand Function in Breast Cancer Survivors
Brief Title: The Effect of Hand Exercises on Upper Limb Volume, Quality of Life, and Hand Function in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Presbyterian Healthcare Services (Unknown)
Responsible Party: Principal Investigator, Elisabeth Wise, Primary Investigator, Physical Therapist, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FY2023-183
Record Dates: First submitted 2023-07-20; First posted 2023-08-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Two groups will be compared, with treatment occurring at the same time. One group will receive the experimental exercises plus the usual treatment, the comparison group will only receive the usual treatment for breast cancer-related lymphedema.
Who Masked: Participant
Masking Description: Participants will be masked regarding whether they are assigned to the intervention or comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will receive hand mobility and grip strengthening exercises in addition to the usual care for breast cancer-related lymphedema of the upper limb.
  Interventions: Other: Hand Mobility and Grip Strengthening Exercises; Other: Usual Care
- Comparison (Active Comparator): Participants will receive only the usual care for breast cancer-related lymphedema.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Hand Mobility and Grip Strengthening Exercises — Addition of hand mobility and grip strengthening exercises to the usual care for breast cancer-related lymphedema to assess changes in limb volume, quality of life, and hand function.
  Arms: Experimental
Other: Usual Care — Manual lymphatic drainage, compression, exercise, skin hygiene.

SUMMARY:
The purpose of this study is to determine whether the addition of simple hand mobility and grip strengthening exercises to the usual care for upper extremity lymphedema will reduce limb volume and improve the quality of life, hand dexterity, and grip strength for those experiencing breast cancer-related lymphedema. Researchers will compare those receiving the usual treatment to those receiving the usual treatment plus hand mobility and grip strengthening exercises.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the addition of simple hand mobility and grip strengthening exercises to the usual care for upper extremity lymphedema will reduce limb volume and improve the quality of life, hand dexterity, and grip strength for those experiencing early, moderate, or late stage breast cancer-related lymphedema.

This study is an experimental clinical trial to determine the effectiveness of hand mobility and grip exercises on limb volume, quality of life, hand dexterity, and grip strength in women with breast cancer-related lymphedema. The two independent variables are group, a between-subject factor, and time, a within subject factor. There are two levels of the independent variable of group: (1)usual care plus hand exercises and (2) usual care alone. The independent variable of time will be assessed at three timepoints: initial to 4 weeks, 4 to 8 weeks, and initial to 8 weeks of intervention. The four dependent variables are: (1) upper limb volume, (2) quality of life, (3) hand dexterity, and (4) grip strength. If a relationship (r>0.5) is found between any of the dependent variables, MANOVA will used for analysis. If no relationship is found, a 2x3 mixed ANOVA will be used to analyze each dependent variable without a significant relationship to the others. The comparison group will receive the usual physical or occupational therapy treatment, including compression bandaging, manual lymphatic drainage, shoulder and scapular muscle exercises, and education regarding skin hygiene and monitoring. The experimental group will receive the usual treatment plus additional hand mobility and grip strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* Biologic women age 18 years or older with a diagnosis of clinical lymphedema of one upper extremity-early (clinical), moderate, or late stage, following treatment for breast cancer within the previous 10 years.
* Women concurrently receiving immunotherapy or chemotherapy are eligible for inclusion, but an additional information request may be necessary (e.g., any activity restrictions and nadir periods) to determine whether they can safely participate in the exercise activities and apply compression.

Exclusion Criteria:

* Prior history of paresis in either upper limb, though paresis related to nerve compression from increased lymphatic volume will be eligible for inclusion.
* Current open wounds (> 0.5 inch in length or diameter) of the axilla or edematous upper limb would be excluded, though the presence of lymphorrhea without visible skin tears will be eligible for inclusion.
* Previous treatment for upper limb lymphedema or a prior diagnosis of congestive heart failure or end-stage renal disease due to the impact on edematous limbs and risk of cardiac overload.
* Women who cannot speak or read English or Spanish sufficiently to complete the Lymphedema Life Impact Scale or understand the consent forms, educational information, and printed exercises will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologic women due to increased prevalence of breast cancer diagnosis.
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Upper Limb volume | Day 1, at 4 weeks, at 8 weeks of treatment/completion of study.
  Circumferential measurements of the upper limb, converted to volumetric measurements with frustrum equation through Epic EMR.

SECONDARY OUTCOMES:
Grip Strength | Day 1, at 4 weeks, and at 8 weeks of treatment/completion of study.
  Grip Strength assessed with Jamar Hand Dynamometer.
Nine-Hole Peg Test | Day 1, at 4 weeks, and at 8 weeks of treatment/completion of study.
  Nine-Hole Peg Test with affected limb only to assess dexterity.
Lymphedema Life Impact Scale | Day 1, at 4 weeks, and at 8 weeks of treatment/completion of study.
  Participants fill out Lymphedema Life Impact Scale, a self-report survey to assess quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Wise, DPT, Principal Investigator — Texas Woman's University
Locations (3):
- United States (3):
  - Presbyterian Healthplex, Albuquerque, New Mexico
  - Presbyterian Southern Outpatient Rehab, Rio Rancho, New Mexico
  - Presbyterian Santa Fe Medical Center, Santa Fe, New Mexico

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Background] Ahmad FB, Anderson RN. The Leading Causes of Death in the US for 2020. JAMA. 2021 May 11;325(18):1829-1830. doi: 10.1001/jama.2021.5469. No abstract available. PMID 33787821
- [Background] Ahmed RL, Prizment A, Lazovich D, Schmitz KH, Folsom AR. Lymphedema and quality of life in breast cancer survivors: the Iowa Women's Health Study. J Clin Oncol. 2008 Dec 10;26(35):5689-96. doi: 10.1200/JCO.2008.16.4731. Epub 2008 Nov 10. PMID 19001331
- [Background] Chromy A, Zalud L, Dobsak P, Suskevic I, Mrkvicova V. Limb volume measurements: comparison of accuracy and decisive parameters of the most used present methods. Springerplus. 2015 Nov 19;4:707. doi: 10.1186/s40064-015-1468-7. eCollection 2015. PMID 26618096
- [Background] Davies C, Levenhagen K, Ryans K, Perdomo M, Gilchrist L. Interventions for Breast Cancer-Related Lymphedema: Clinical Practice Guideline From the Academy of Oncologic Physical Therapy of APTA. Phys Ther. 2020 Jul 19;100(7):1163-1179. doi: 10.1093/ptj/pzaa087. PMID 32589208
- [Background] De Groef A, Van Kampen M, Dieltjens E, Christiaens MR, Neven P, Geraerts I, Devoogdt N. Effectiveness of postoperative physical therapy for upper-limb impairments after breast cancer treatment: a systematic review. Arch Phys Med Rehabil. 2015 Jun;96(6):1140-53. doi: 10.1016/j.apmr.2015.01.006. Epub 2015 Jan 13. PMID 25595999
- [Background] Feys P, Lamers I, Francis G, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. The Nine-Hole Peg Test as a manual dexterity performance measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):711-720. doi: 10.1177/1352458517690824. Epub 2017 Feb 16. PMID 28206826
- [Background] Giray E, Akyuz G. Assessment of Family Caregiver Burden and Its Relationships Between Quality of Life, Arm Disability, Grip Strength, and Lymphedema Symptoms in Women with Postmastectomy Lymphedema: A Prospective Cross-Sectional Study. Eur J Breast Health. 2019 Feb 15;15(2):111-118. doi: 10.5152/ejbh.2019.4385. eCollection 2019 Apr. PMID 31001613

DOCUMENTS (1):
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT05983380/ICF_000.pdf